CLINICAL TRIAL: NCT06465251
Title: Effects of Repetition Home-based Constraint Induced Movement Therapy (CIMT) Compared With Repetition Clinic-based CIMT on Outcomes Post Stroke: A Randomized Controlled Trial
Brief Title: Effects of Home-based CIMT and Clinic-based CIM on Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Shamay Ng, Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-CIMT
Record Dates: First submitted 2024-06-13; First posted 2024-06-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Motor Function
Keywords: Constraint Induced Movement Therapy; Disability

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home-based CIMT (Experimental): Participants and their families will be required to attend clinic to practice 3 times (Monday, Wednesday and Friday) during the first week, 2 times (Monday and Friday) during the second week and once (Monday) during the 3rd week under the supervision of a trained research assistant. They will be allowed to practice exclusively at home during the 4th week under the supervision of their family members.
  Interventions: Device: Home-based CIMT
- Clinic-based CIMT (Experimental): Participants in both groups will perform 5 tasks with the affected upper limb, each 100 times, making it 500 repetitions in total within a duration of 2 hours every day, five days a week for 4 weeks at home and in the clinic respectively. Details of the tasks to be performed are presented in table 1. We chose 2 hours because, patients with stroke can perform about 300 repetitions of tasks practice within one hour (Birkinmeier et al., 2014). Similarly, we chose 500 repetitions because the number of repetitions of tasks practice required for motor recovery ranges between 300 and 600 repetitions per day
  Interventions: Device: Clinic-based CIMT
- Control (Placebo Comparator): Participants will attend 45 minutes health talk provided by a research assistant twice in a week (Mondays and Fridays) in the clinic for 4 weeks. They will receive each talk in either a group of 3 or 5 patients. Similar control intervention was used in previous study
  Interventions: Device: Control

INTERVENTIONS:
Device: Home-based CIMT — Participants and their families will be required to attend clinic to practice 3 times (Monday, Wednesday and Friday) during the first week, 2 times (Monday and Friday) during the second week and once (Monday) during the 3rd week under the supervision of a trained research assistant. They will be allowed to practice exclusively at home during the 4th week under the supervision of their family members.
  Arms: Home-based CIMT
Device: Clinic-based CIMT — Participants in both groups will perform 5 tasks with the affected upper limb, each 100 times, making it 500 repetitions in total within a duration of 2 hours every day, five days a week for 4 weeks at home and in the clinic respectively. Details of the tasks to be performed are presented in table 1. We chose 2 hours because, patients with stroke can perform about 300 repetitions of tasks practice within one hour. Similarly, we chose 500 repetitions because the number of repetitions of tasks practice required for motor recovery ranges between 300 and 600 repetitions per day
  Arms: Clinic-based CIMT
Device: Control — Participants will attend 45 minutes health talk provided by a research assistant twice in a week (Mondays and Fridays) in the clinic for 4 weeks. They will receive each talk in either a group of 3 or 5 patients. Similar control intervention was used in previous study
  Arms: Control

SUMMARY:
Constraint induced movement therapy (CIMT) is based on the theoretical basis that constraining the unaffected limb following injury of the brain such as stroke can help overcome learned non-use. It comprises of constraint of the unaffected limb, massed tasks practice with the affected limb and a behavioral contract known as the transfer package whereby use of the affected limb is extended to the real-world situations. home-based rehabilitation is likely to be cost-effective, and it may reduce cost for patients in terms of hospital charges and transport fares. However, one of the major problems with the existing home-based CIMT protocols is that, they used number of hours spent carrying out tasks practice as the measure of intensity of practice, and it has been argued that, such method is not clear and it does not reflect the correct intensity of practice.

DETAILED DESCRIPTION:
The aim of this study is to determine the effects of home-based CIMT compared with clinic-based CIMT that use number of repetition of tasks practice on motor impairment, motor function, quantity and quality of use of the limb in everyday life, community integration, stroke self-efficacy and quality of life. Constraint induced movement therapy (CIMT) can be administered either at home or in the clinic. The home-based CIMT is used to make CIMT easier for the patients

ELIGIBILITY:
Inclusion Criteria:

* have stroke 1-2 years before
* moderate disability
* a score of 1 to 3 on the motor arm item of the National Institutes of Health Stroke Scale (NIHSS)
* a score of 3 or more on the upper arm item of the Motor Assessment Scale (MAS)
* no significant cognitive impairment (a score of ≥24 points on Minimental state examination)

Exclusion Criteria:

* patients with re-stroke
* serious orthopaedic conditions such joint contracture, osteoarthritis and burns that will interfere with carrying out CIMT
* who are receiving rehabilitation at the time of the study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
upper limb Fugl Meyer motor assessment | at baseline
  valid and reliable instrument that assesses motor impairment following stroke. Items in the instrument are scored on a scale between 0 and 2, with a score 0 indicating cannot perform, a score of 1 indicating performs partially, and a score of 2 indicating performs fully. Scores obtained from the instrument can range from 0 to 66, with higher scores denoting higher ability.
upper limb Fugl Meyer motor assessment | 2 weeks
  valid and reliable instrument that assesses motor impairment following stroke . Items in the instrument are scored on a scale between 0 and 2, with a score 0 indicating cannot perform, a score of 1 indicating performs partially, and a score of 2 indicating performs fully. Scores obtained from the instrument can range from 0 to 66, with higher scores denoting higher ability.
upper limb Fugl Meyer motor assessment | 4 weeks
  valid and reliable instrument that assesses motor impairment following stroke. Items in the instrument are scored on a scale between 0 and 2, with a score 0 indicating cannot perform, a score of 1 indicating performs partially, and a score of 2 indicating performs fully. Scores obtained from the instrument can range from 0 to 66, with higher scores denoting higher ability.
upper limb Fugl Meyer motor assessment | 3 months follow up
  valid and reliable instrument that assesses motor impairment following stroke . Items in the instrument are scored on a scale between 0 and 2, with a score 0 indicating cannot perform, a score of 1 indicating performs partially, and a score of 2 indicating performs fully. Scores obtained from the instrument can range from 0 to 66, with higher scores denoting higher ability.
Wolf motor function test (WMFT) | at baseline
  valid and reliable tool comprising of 17 items that assess motor function of the upper limb following stroke. Each of the items is rated on a scale of zero to 5, with higher scores denoting higher motor function. Similarly, the MAL is a valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
Wolf motor function test (WMFT) | 2 weeks
  valid and reliable tool comprising of 17 items that assess motor function of the upper limb following stroke. Each of the items is rated on a scale of zero to 5, with higher scores denoting higher motor function. Similarly, the MAL is a valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
Wolf motor function test (WMFT) | 4 weeks
  valid and reliable tool comprising of 17 items that assess motor function of the upper limb following stroke. Each of the items is rated on a scale of zero to 5, with higher scores denoting higher motor function. Similarly, the MAL is a valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
Wolf motor function test (WMFT) | 3 months follow up
  valid and reliable tool comprising of 17 items that assess motor function of the upper limb following stroke. Each of the items is rated on a scale of zero to 5, with higher scores denoting higher motor function. Similarly, the MAL is a valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
motor activity log (MAL) | At baseline
  valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
motor activity log (MAL) | 2 weeks
  valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
motor activity log (MAL) | 4 weeks
  valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
motor activity log (MAL) | 3 months follow up
  valid and reliable instrument comprising of 30 items that separately assess quantity and quality of the use of upper extremity in real world following a stroke. Each of the items contained in the instrument are rated on a scale of zero to 5, with higher scores denoting higher quantity or quality of use of the limb in the real world.
community integration measure (CIM) | at baseline
  valid and reliable 10-item measure of social interactions following a disease or illness. Each item is rated on a 5 point scale, with possible scores ranging from 0 to 50.
community integration measure (CIM) | 2 weeks
  valid and reliable 10-item measure of social interactions following a disease or illness. Each item is rated on a 5 point scale, with possible scores ranging from 0 to 50.
community integration measure (CIM) | 4 weeks
  valid and reliable 10-item measure of social interactions following a disease or illness. Each item is rated on a 5 point scale, with possible scores ranging from 0 to 50.
community integration measure (CIM) | 3 months follow up
  valid and reliable 10-item measure of social interactions following a disease or illness. Each item is rated on a 5 point scale, with possible scores ranging from 0 to 50.
stroke self-efficacy questionnaire (SSEQ) | at baseline
  The SSEQ is a valid and reliable measure of how confident patients with stroke are in carrying out activities of daily living. The most recent version of the questionnaire is scored on a scale of 0 to 3, with higher scores denoting increasing confidence.
stroke self-efficacy questionnaire (SSEQ) | 2 weeks
  The SSEQ is a valid and reliable measure of how confident patients with stroke are in carrying out activities of daily living. The most recent version of the questionnaire is scored on a scale of 0 to 3, with higher scores denoting increasing confidence.
stroke self-efficacy questionnaire (SSEQ) | 4 weeks
  The SSEQ is a valid and reliable measure of how confident patients with stroke are in carrying out activities of daily living. The most recent version of the questionnaire is scored on a scale of 0 to 3, with higher scores denoting increasing confidence.
stroke self-efficacy questionnaire (SSEQ) | 3 months follow up
  The SSEQ is a valid and reliable measure of how confident patients with stroke are in carrying out activities of daily living. The most recent version of the questionnaire is scored on a scale of 0 to 3, with higher scores denoting increasing confidence.
stroke specific quality of life (SSQoL) | at baseline
  valid and reliable measure of quality of life specifically for patients with stroke. It consists of 49 items measuring 12 domains.
stroke specific quality of life (SSQoL) | 2 weeks
  valid and reliable measure of quality of life specifically for patients with stroke. It consists of 49 items measuring 12 domains.
stroke specific quality of life (SSQoL) | 4 weeks
  valid and reliable measure of quality of life specifically for patients with stroke. It consists of 49 items measuring 12 domains.
stroke specific quality of life (SSQoL) | 3 months follow up
  valid and reliable measure of quality of life specifically for patients with stroke. It consists of 49 items measuring 12 domains.

CONTACTS AND LOCATIONS:
Overall Officials: Shamay Ng, PhD, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong